CLINICAL TRIAL: NCT04634149
Title: An Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-986036 in Participants With Normal Hepatic Function and Participants With Moderate and Severe Hepatic Impairment
Brief Title: A Study to Evaluate the Drug Levels, Safety, and Tolerability of BMS-986036 in Participants With Normal Liver Function and Participants With Moderate and Severe Liver Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB130-112
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Moderate Liver Impairment; Severe Liver Impairment
Keywords: Cirrhosis; Hepatic impairment; Liver impairment; Nonalcoholic steatohepatitis (NASH)
MeSH Terms: conditions — Fibrosis; Non-alcoholic Fatty Liver Disease | interventions — Pegbelfermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A: Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: BMS-986036
- Group B: Severe Hepatic Impairment (Experimental)
  Interventions: Drug: BMS-986036
- Group C: Normal Hepatic Function (Experimental)
  Interventions: Drug: BMS-986036

INTERVENTIONS:
Drug: BMS-986036 — Specified dose on specified days

SUMMARY:
The purpose of this study is to investigate the effect of impaired liver function on the drug levels, safety, and tolerability of BMS-986036 in participants with moderate and severe liver impairment. Results from this study will be used to determine whether dose adjustment is required for patients with decreased liver function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants or participants with hepatic impairment, as determined by medical history, physical exam, electrocardiogram (ECG), and clinical laboratory determinations
* Body mass index (BMI) of 18.0 kg/m^2 to 40.0 kg/m^2, inclusive. BMI = weight (kg)/height (m^2)

Exclusion Criteria:

* Any history of known or suspected congenital or acquired immunodeficiency state or condition that would have compromised the participant's immune status
* History of biliary disorders, including Gilbert's syndrome or Dubin-Johnson disease

Other protocol-defined inclusion/exclusion criteria apply

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 29 days
Time of maximum observed plasma concentration (Tmax) | Up to 29 days
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC(0-T)) | Up to 29 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 31 days
Number of participants with clinical laboratory abnormalities | Up to 31 days
Number of participants with vital sign abnormalities | Up to 31 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 31 days
Number of participants with physical examination abnormalities | Up to 31 days
Maximum observed plasma concentration (Cmax) | Up to 29 days
Time of maximum observed plasma concentration (Tmax) | Up to 29 days
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration(AUC(0-T)) | Up to 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution - 0002, Miami, Florida
  - Local Institution, Orlando, Florida
  - Local Institution - 0001, San Antonio, Texas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm